CLINICAL TRIAL: NCT00932802
Title: GIANT - Greatest International Antiinfective Trial With Avelox®
Brief Title: Greatest International Antiinfective Trial With Avelox
Acronym: GIANT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Bayer Schering Pharma AG, Medical Affairs Therapeutic Area Head
Other Study IDs: 12219; AX0401 (Other: Company Internal); 11828 (Other: Company Internal); 12206 (Other: Company Internal); 12214 (Other: Company Internal); 12234 (Other: Company Internal); 12213 (Other: Company Internal); 12212 (Other: Company Internal); 12216 (Other: Company Internal); 12220 (Other: Company Internal); 12219 (Other: Company Internal); 12217 (Other: Company Internal); 12225 (Other: Company Internal); 12223 (Other: Company Internal); 12229 (Other: Company Internal); 12221 (Other: Company Internal); 12218 (Other: Company Internal); 12222 (Other: Company Internal); 12230 (Other: Company Internal); 12211 (Other: Company Internal); 12227 (Other: Company Internal); 12228 (Other: Company Internal); 12226 (Other: Company Internal); 12235 (Other: Company Internal); 12233 (Other: Company Internal); 12224 (Other: Company Internal); 12215 (Other: Company Internal); 12231 (Other: Company Internal); 12232 (Other: Company Internal)
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Bronchitis, Chronic; Bronchial Diseases
Keywords: Non-Interventional; Observational; NIS; Moxifloxacin; MXF; Avelox; AECB
MeSH Terms: conditions — Bronchitis, Chronic; Bronchial Diseases | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — AECB patients under daily life treatment receiving moxifloxacin according to the local product information.

SUMMARY:
The observation period for each patient covered an initial treatment period with Avelox® plus optional 2 long-term follow-up periods (6 and 12 months).For each patient, the physician documented data at any initial visit (baseline) and at least one short-term follow-up visit (=initial treatment period).Optionally, long-term follow-ups (6 and 12 months) were documented, and a patient questionnaire was filled in.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with diagnosis of AECB and decision taken by the investigator to prescribe moxifloxacin

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of AECB who take moxifloxacin
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2004-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of impact of AECB on the patient and the community as well as effect and safety of a treatment with moxifloxacin tablets in daily life clinical practice | During documentation at baseline and at at least one short-term follow-up visit; at maximum two short-term (within ca. 14 days) and two long-term follow-up visits (after ca. 6 and 12 months).

SECONDARY OUTCOMES:
Course of symptom relief | During documentation of up to two short-term follow-up visits (within ca. 14 days)
Speed of return to normal daily life activities | During documentation of the last short-term follow-up visit (after ca. 14 days)
Adverse events collection | Throughout the entire study, whenever Adverse Events occur
Evaluation of frequency of new exacerbations | During documentation of up to two long-term follow-up visits (after ca. 6 and 12 months)
Progression of chronic respiratory disease | During documentation of up to two long-term follow-up visits (after ca. 6 and 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (24):
- Many Locations, Austria
- Many Locations, Brazil
- Many Locations, China
- Many Locations, Colombia
- Many Locations, Croatia
- Many Locations, Egypt
- Many Locations, El Salvador
- Many Locations, Germany
- Many Locations, Hong Kong
- Many Locations, Hungary
- Many Locations, Indonesia
- Many Locations, Malaysia
- Many Locations, Mexico
- Many Locations, Morocco
- Many Locations, Netherlands
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Poland
- Many Locations, Singapore
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Switzerland
- Many Locations, Taiwan
- Many Locations, Turkey (Türkiye)

REFERENCES:
- [Result] Anzueto A, Miravitlles M, Ewig S, Legnani D, Heldner S, Stauch K. Identifying patients at risk of late recovery (>/= 8 days) from acute exacerbation of chronic bronchitis and COPD. Respir Med. 2012 Sep;106(9):1258-67. doi: 10.1016/j.rmed.2012.06.002. Epub 2012 Jun 30. PMID 22749710